CLINICAL TRIAL: NCT07219212
Title: A Study of JNJ-90301900 in Combination With Concurrent Chemoradiation Therapy in Participants With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of JNJ-90301900 in Combination With Chemoradiation Therapy in Participants With Locally Advanced Head and Neck Squamous Cell Carcinoma
Acronym: LUMIRAY
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Enterprise Innovation Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90301900HNC1001; 90301900HNC1001 (Other: Janssen Research & Development, LLC); 2025-522914-22-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-90301900 + Concurrent Chemoradiation Therapy (cCRT) (Experimental): Participants will receive JNJ-90301900 administered intratumorally and/or intranodally, in combination with concurrent chemoradiation therapy (cCRT) consisting of cisplatin and intensity-modulated radiation therapy (IMRT). Post-treatment follow-up will continue until the end of study (EOS), radiographic disease progression, study discontinuation, or study completion, whichever occurs first.
  Interventions: Drug: JNJ-90301900; Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Drug: JNJ-90301900 — JNJ-90301900 will administered via intratumoral and/or intranodal injection.
  Other Names: NBTXR3; Functionalized hafnium oxide nanoparticles
Drug: Cisplatin — Cisplatin will be administered intravenously.
Radiation: Intensity Modulated Radiation Therapy (IMRT) — IMRT radiation therapy will be administered.

SUMMARY:
This global, open-label, single arm, phase 1b study aims to learn more about whether a treatment called JNJ-90301900 is safe and effective when injected directly into tumors, along with standard chemotherapy and radiation therapy, for participants with head and neck squamous cell cancer (HNSCC; a type of solid tumor that begins in outer tissue layer of the mouth & throat).

ELIGIBILITY:
Inclusion criteria:

* Pathologically (histologically or cytologically) proven diagnosis of HNSCC of the oral cavity, oropharynx (p16 negative), hypopharynx, or supraglottic larynx
* Stage III, IVA or IVB according to the 8th Edition of the American Joint Committee on Cancer (AJCC) guidelines
* A candidate for definitive concurrent chemoradiation therapy treatment as determined by investigator and per local guidelines
* Participants must have at least 1 target lesion (primary tumor or involved lymph node) per RECIST v.1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1

Exclusion criteria:

* Primary tumor originating in the nasopharynx, paranasal sinuses, salivary glands, thyroid gland, parathyroid gland, skin, or unknown primary site
* Non-squamous histology
* Stages 0, I, II, and IVC HNSCC, loco-regionally recurrent HNSCC, or synchronous second primary HNSCC (within 2 months)
* Ineligible to receive cisplatin chemotherapy
* Suspected or known allergies, hypersensitivity, or intolerance to JNJ-90301900 or its excipients

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2028-07-14 (Estimated); Study Completion 2028-07-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) by Severity | Up to approximately 2 years 14 weeks
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v) 5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) According to RECIST v.1.1 | Up to approximately 2 years 14 weeks
  ORR defined as percentage of participants achieving complete response (CR) or partial response (PR) by investigator assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
Complete Response (CR) Rate | Up to approximately 2 years 12 weeks
  Percentage of participants achieving CR according to RECIST v.1.1 will be reported.
Disease Control Rate (DCR) | Up to approximately 2 years 12 weeks
  DCR is defined as the percentage of participants achieving CR, PR, or stable disease (SD) as per RECIST v.1.1 criteria.
Injected Tumor Response Rate | Up to approximately 2 years 14 weeks
  Response rate will be measured based on total tumor shrinkage compared to baseline among those lesions injected with JNJ-90301900.
Time to Locoregional Failure (LRF) | Up to approximately 2 years 14 weeks
  Time to LRF is defined as time from enrollment to first failure of LRF using investigator RECIST v.1.1 assessments.
Time to Distant Failure (DF) | Up to approximately 2 years 14 weeks
  Time to DF is defined as time from enrollment to first failure of DF using investigator RECIST v.1.1 assessments.
Progression Free Survival (PFS) | Up to approximately 2 years 14 weeks
  PFS is defined as the time from enrollment to radiographic disease progression, or death from any cause, whichever occurs first.
Number of Participants with Post-Radiation Neck Dissection (PRND) | Up to approximately 2 years 14 weeks
  Participants with PRND will be summarized and will continue to be radiographically evaluated for response by RECIST v.1.1.
Number of Participants with Post-Radiation Primary Salvage Surgery | Up to approximately 2 years 14 weeks
  Participants with post-radiation primary salvage surgery will be summarized and will continue to be radiographically evaluated for response by RECIST v.1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Enterprise Innovation, Inc. Clinical Trial, Study Director — Johnson & Johnson Enterprise Innovation Inc.
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Emory University, Atlanta, Georgia
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency